CLINICAL TRIAL: NCT03701763
Title: A PHASE 3, MULTI-CENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO ASSESS THE EFFICACY AND SAFETY OF APREMILAST (CC-10004) IN PEDIATRIC SUBJECTS FROM 6 THROUGH 17 YEARS WITH MODERATE TO SEVERE PLAQUE PSORIASIS
Brief Title: Efficacy and Safety Study of Apremilast (CC-10004) in Pediatric Subjects From 6 Through 17 Years of Age With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PPSO-003; U1111-1219-3112 (Registry Identifier: WHO); 2018-002918-12 (EudraCT Number)
Expanded Access: NCT03740516 (No longer available)
Record Dates: First submitted 2018-08-30; First posted 2018-10-10 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Psoriasis
Keywords: Pediatric; 6 through 17 years; Plaque Psoriasis; Psoriasis; CC-10004; Apremilast; Otezla; Children; Adolescents; SPROUT
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Administration of Apremilast (CC-10004) - 20mg (Experimental): Apremilast 20mg Twice Daily (BID)
  Interventions: Drug: Apremilast (CC-10004)
- Administration of Apremilast (CC-10004) - 30mg (Experimental): Apremilast 30mg Twice Daily (BID)
  Interventions: Drug: Apremilast (CC-10004)
- Administration of Placebo (Placebo Comparator): Placebo tablet Twice Daily (BID)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Apremilast (CC-10004) — Apremilast (CC-10004)
  Arms: Administration of Apremilast (CC-10004) - 20mg; Administration of Apremilast (CC-10004) - 30mg
Other: Placebo — Placebo
  Arms: Administration of Placebo

SUMMARY:
This is a Phase 3, multicenter, randomized, placebo-controlled, double-blind study of the efficacy and safety of apremilast (CC-10004) in pediatric subjects with moderate to severe plaque psoriasis.

At least 230 pediatric subjects (ages 6 through 17 years) will be randomized 2:1 to receive either apremilast or placebo for the first 16 weeks and then all subjects will receive apremilast during the 36 week Extension Phase for a total of 52 weeks. Randomization to apremilast arm or placebo arm will be stratified by age group (6 to 11 years or 12 to 17 years). Subjects will receive apremilast treatment of either 20 mg twice daily (BID) or 30 mg BID, depending on weight. This Phase 3 study is being conducted to evaluate the safety and efficacy of apremilast in the treatment of pediatric subjects.

DETAILED DESCRIPTION:
Treatment will be assigned by weight with subjects 20 kg to < 50 kg receiving apremilast 20 mg BID or placebo BID and subjects ≥ 50 kg receiving apremilast 30 mg BID or placebo BID. Total study duration is up to 71 weeks. Subjects completing all 52 weeks of the treatment and extension phase will be able to enter the Long-term study. Subjects not entering the Long-term study will return for 3 observational follow-up visits, 4, 8 and 14 weeks after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Males or female subjects 6 to 17 years of age, inclusive, at the time the informed consent form is signed by the legal guardian
2. Subjects must have a weight of ≥ 20 kg
3. Diagnosis of chronic plaque psoriasis for at least 6 months prior to Screening.
4. Has moderate to severe plaque psoriasis at Screening and Baseline as defined by:

   * PASI score ≥ 12; and
   * Body surface area (BSA) ≥ 10%; and
   * sPGA ≥ 3 (moderate to severe)
5. Disease inadequately controlled by or inappropriate for topical therapy for psoriasis
6. Candidate for systemic therapy or phototherapy

Exclusion Criteria:

1. Guttate, erythrodermic, or pustular psoriasis at Screening and Baseline
2. Psoriasis flare or rebound within 4 weeks prior to Screening
3. Prior history of suicide attempt at any time in the subject's lifetime prior to Screening or randomization in the study, or major psychiatric illness requiring hospitalization within 3 years prior to signing the assent and informed consent
4. Answer "Yes" to any question on the Columbia-Suicide Severity Rating Scale during Screening or at Baseline
5. Current or planned concurrent use of the following therapies that may have a possible effect on psoriasis

   a. Topical therapy within 2 weeks prior to randomization (including but not limited to topical corticosteroids, topical retinoid or vitamin D analog preparations, tacrolimus, pimecrolimus, or anthralin/dithranol)

   Exceptions*:

   i. Low potency or weak corticosteroids (please refer to the Investigators' Manual) will be allowed as background therapy for treatment of the face, axillae and groin in accordance with manufacturer's suggested usage ii. Unmedicated skin moisturizer (eg, Eucerin®) will also be permitted for body lesions

   *Subjects should not use these topical treatments within 24 hours prior to the clinic visit.

   b. Conventional systemic therapy for psoriasis within 4 weeks prior to randomization c. Phototherapy treatment (ie, ultraviolet B [UVB], PUVA) within 4 weeks prior to randomization d. Biologic therapy within 4 weeks prior to randomization or 5 PK/PD half-lives (whichever is longer).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 245 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (99):
- United States (39):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Johnson Dermatology Clinic, Fort Smith, Arkansas
  - Zenith Research Inc., Beverly Hills, California
  - First OC Dermatology, Fountain Valley, California
  - Avance Clinical Trials, Laguna Niguel, California
  - Stanford University, Palo Alto, California
  - Coastal Family Dermatology, San Luis Obispo, California
  - University of California Los Angeles, Santa Monica, California
  - California Dermatology Institute, Thousand Oaks, California
  - Solutions Through Advanced Research Inc, Jacksonville, Florida
  - Glick Skin Institute Clinical Research, Margate, Florida
  - University of Miami Hospital, Miami, Florida
  - Ciocca Dermatology, Miami, Florida
  - University of South Florida Health Morsani Center for Advanced Healthcare, Tampa, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Treasure Valley Medical Research, Meridian, Idaho
  - DeNova Research, Chicago, Illinois
  - Dawes Fretzin Dermatology Group Inc, Indianapolis, Indiana
  - Epiphany Dermatology of Kansas, LLC, Overland Park, Kansas
  - ActivMed Practices and Research Inc, Beverly, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - J Woodson Dermatology and Associates Ltd, Henderson, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Forest Hills Dermatology Group, Forest Hills, New York
  - SUNY Downstate Medical Center, Manhasset, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Essential Medical Research, LLC, Tulsa, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Arlington Research Center, Arlington, Texas
  - Driscoll Childrens Hospital, Corpus Christi, Texas
  - Modern Research Associates PLLC, Dallas, Texas
  - Mosaic Dermatology, Houston, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Jordan Valley Dermatology Center, West Jordan, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - Centre Hospitalier Universitaire Saint Pierre, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Canada (7):
  - Kirk Barber Research, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Enverus Medical Research, Surrey, British Columbia
  - Winnipeg Clinic Dermatology Research, Winnipeg, Manitoba
  - Karma Clinical Trials, St. John's, Newfoundland and Labrador
  - AvantDerm, Toronto, Ontario
  - CHU Saint-Justine, Montreal, Quebec
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Synexus Czech sro, Prague
- France (10):
  - Centre Hospitalier Victor Dupouy Argenteuil, Argenteuil
  - Centre Hospitalier Universitaire Lyon, Bron
  - Cabinet du Docteur Ruer-Mulard Mireille, Martigues
  - Hotel Dieu CHU Nantes, Nantes
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hopital Necker, Paris
  - Centre Hospitalier de Cornouaille - Hopital Laennec, Quimper
  - CHU Saint Etienne Hopital Nord, Saint-Priest En Jarrez
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
  - Centre Hospitalier de Valence, Valence
- Chaim Sheba Medical Center, Ramat Gan, Israel
- Italy (8):
  - Azienda Ospedaliero Universitaria Di Bologna Policlinico S Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria di Cagliari, Cagliari
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera di Reggio Emilia Arcispedale Santa Maria Nuova, Reggio Emilia
  - Policlinico Tor Vergata, Roma
  - Istituto Dermatologico San Gallicano IRCCS Dermatologia Clinica, Roma
- Radboud university medical center, Nijmegen, Netherlands
- Russia (15):
  - Altai State Medical University, Barnaul
  - Chelyabinsk Regional Clinical Skin and Venereal Dispensary, Chelyabinsk
  - Republican Clinical Dermatology and Venerology Dispensary, Kazan'
  - Clinical Dispensary of Dermatology and Venereology of Krasnodar Territory of the Ministry of Health, Krasnodar
  - State Scientific Center for Dermatovenereology and Cosmetology, Moscow
  - Russian Children's Clinical Hospital, Moscow
  - Moscow Scientific Practical Center of Dermatology Venerology and Cosmetology, Moscow
  - National Medical Research Center for Children's Health, Moscow
  - LLC Medical Center Zdorovaya Semiya, Novosibirsk
  - Pierre Wolkenshtein Skin Diseases Clinic LLC, Saint Petersburg
  - LLC PiterKlinika, Saint Petersburg
  - Saint Petersburg State Pediatric Medical University, Saint Petesburg
  - Bashkiria State Medical University, Ufa
  - Yarosavl State Medical Academy, Yaroslavl
  - Ural Scientific Research Institute of Dermatovenereology and Immunopathology, Yekaterinburg
- Spain (12):
  - Hospital Marques de Valdecilla, Santander, Cantabria
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital Universitari Germans Trias i Pujol Can Ruti, Badalona
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Complexo Hospitalario De Pontevedra, Pontevedra
  - Hospital Universitario Virgen del Rocio - PPDS, Seville

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Fiorillo L, Becker E, de Lucas R, Belloni-Fortina A, Armesto S, Elewski B, Maes P, Oberoi RK, Paris M, Zhang W, Zhang Z, Arkin L. Efficacy and safety of apremilast in pediatric patients with moderate-to-severe plaque psoriasis: 16-week results from SPROUT, a randomized controlled trial. J Am Acad Dermatol. 2024 Jun;90(6):1232-1239. doi: 10.1016/j.jaad.2023.11.068. Epub 2024 Jan 23. PMID 38266683
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into this study at sites in Belgium, Canada, Czech Republic, France, Israel, Italy, Russia, Spain, and the United States.
Pre-assignment Details: Screening tests and procedures were performed up to 35 days preceding randomization.
Groups:
- Placebo: In the placebo-controlled phase, participants who were randomized to placebo received placebo twice daily (BID) for 16 weeks. At Week 16, participants in the placebo group were switched to apremilast based on baseline weight. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Apremilast: In the placebo-controlled phase, participants who were randomized to apremilast who were 20 to < 50 kg received apremilast 20 mg twice daily (BID) for 16 weeks, and participants >/= 50 kg received apremilast 30 mg BID for 16 weeks. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Placebo/Apremilast: At Week 16, participants in the placebo group during the placebo-controlled phase were switched to apremilast based on baseline weight. Participants 20 to < 50 kg received apremilast 20 mg BID for 36 weeks, and participants >/= 50 kg received apremilast 30 mg BID for 36 weeks during the apremilast-extension phase. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Apremilast/Apremilast: At Week 16, participants in the apremilast group during the placebo-controlled phase continued to receive their original dosing assignment for an additional 36 weeks during the apremilast-extension phase. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
Period: Placebo-controlled Phase
Arm/Group | Placebo | Apremilast | Placebo/Apremilast | Apremilast/Apremilast
Started | 82 | 163 | 0 (This arm was not included in the Placebo-controlled Phase.) | 0 (This arm was not included in the Placebo-controlled Phase.)
Took at Least 1 Dose of Investigational Product (IP) | 80 | 163 | 0 (This arm was not included in the Placebo-controlled Phase.) | 0 (This arm was not included in the Placebo-controlled Phase.)
Completed | 72 | 149 | 0 (This arm was not included in the Placebo-controlled Phase.) | 0 (This arm was not included in the Placebo-controlled Phase.)
Not Completed | 10 | 14 | 0 | 0
Not completed — Adverse Event | 1 | 5 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0
Not completed — Miscellaneous | 2 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 3 | 5 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0
Period: Apremilast Extension Phase
Arm/Group | Placebo | Apremilast | Placebo/Apremilast | Apremilast/Apremilast
Started | 0 (This arm was not included in the Apremilast Extension Phase.) | 0 (This arm was not included in the Apremilast Extension Phase.) | 72 | 149
Received Apremilast 20mg BID in Either Placebo-controlled or Apremilast Extension Phases (Week 0-52) | 0 (This arm was not included in the Apremilast Extension Phase.) | 0 (This arm was not included in the Apremilast Extension Phase.) | 36 | 80
Received Apremilast 30mg BID in Either Placebo-controlled or Apremilast Extension Phases (Week 0-52) | 0 (This arm was not included in the Apremilast Extension Phase.) | 0 (This arm was not included in the Apremilast Extension Phase.) | 36 | 83
Took at Least 1 Dose of IP | 0 (This arm was not included in the Apremilast Extension Phase.) | 0 (This arm was not included in the Apremilast Extension Phase.) | 72 | 149
Completed | 0 (This arm was not included in the Apremilast Extension Phase.) | 0 (This arm was not included in the Apremilast Extension Phase.) | 61 | 125
Not Completed | 0 | 0 | 11 | 24
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 3 | 8
Not completed — Adverse Event | 0 | 0 | 3 | 1
Not completed — Miscellaneous | 0 | 0 | 2 | 1
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 1 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Non-compliance with Study Drug | 0 | 0 | 1 | 1
Period: 14-Week Observational Follow-up Phase
Arm/Group | Placebo | Apremilast | Placebo/Apremilast | Apremilast/Apremilast
Started | 1 | 4 | 14 | 26
Completed | 1 | 3 | 11 | 23
Not Completed | 0 | 1 | 3 | 3
Not completed — Miscellaneous | 0 | 0 | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Measured in the intent-to-treat (ITT) population, which included all participants who were randomized.
Groups:
- Placebo: In the placebo-controlled phase, participants who were randomized to placebo received placebo twice daily (BID) for 16 weeks. At Week 16, participants in the placebo group were switched to apremilast based on baseline weight. Participants 20 to < 50 kg received apremilast 20 mg BID for 36 weeks, and participants >/= 50 kg received apremilast 30 mg BID for 36 weeks during the apremilast-extension phase. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Apremilast: In the placebo-controlled phase, participants who were randomized to apremilast who were 20 to < 50 kg received apremilast 20 mg twice daily (BID) for 16 weeks, and participants >/= 50 kg received apremilast 30 mg BID for 16 weeks. At Week 16, participants in the apremilast group continued to receive their original dosing assignment for an additional 36 weeks during the apremilast-extension phase. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast | Total
Number analyzed (Participants) | 82 | 163 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (3.25) | 12.3 (3.32) | 12.2 (3.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 89 | 128
  Male | 43 | 74 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 24 | 32
  Not Hispanic or Latino | 71 | 129 | 200
  Unknown or Not Reported | 3 | 10 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 73 | 140 | 213
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) Response at Week 16
Description: The sPGA is the assessment by the Investigator of the overall disease severity of plaque psoriasis at the time of evaluation. The sPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), incorporating an assessment of the severity of the three primary signs of the disease: erythema, scaling and plaque elevation. The results presented are for the percentage of participants with a sPGA response. An sPGA response was defined as a score of clear (0) or almost clear (1) with at least a 2-point reduction from baseline at Week 16.
Time Frame: Baseline to Week 16
Population: Measured in the intent-to-treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 82 | 163
percentage of participants | 11.5 | 33.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Percentage Adjusted Difference = 21.7, 95% CI 2-sided [11.2 to 32.1]

2. Secondary Outcome: Percentage of Participants Who Achieved At Least 75% Reduction in Psoriasis Area Severity Index (PASI-75) From Baseline at Week 16
Description: The Psoriasis Area Severity Index (PASI) is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. The PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. The results presented are for the percentage of participants with PASI-75. PASI-75 was defined as at least a 75% reduction in PASI score from baseline.
Time Frame: Baseline and Week 16
Population: Measured in the intent-to-treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 82 | 163
percentage of participants | 16.1 | 45.4
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Percentage Adjusted Difference = 29.4, 95% CI 2-sided [17.8 to 40.9]

3. Secondary Outcome: Percentage of Participants Who Achieved At Least 50% Reduction in Psoriasis Area Severity Index (PASI-50) From Baseline at Week 16
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. The PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. The results presented are for the percentage of participants with PASI-50. PASI-50 was defined as at least a 50% reduction in PASI score from baseline.
Time Frame: Baseline and Week 16
Population: Measured in the intent-to-treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 82 | 163
percentage of participants | 32.1 | 70.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Percentage Adjusted Difference = 38.4, 95% CI 2-sided [25.6 to 51.2]

4. Secondary Outcome: Percentage Change From Baseline in Total PASI Score at Week 16
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. The PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Positive percentage change from baseline scores indicate a worsening of disease severity, and negative percentage change from baseline scores indicate an improvement in disease severity.
Time Frame: Baseline and Week 16
Population: Measured in the intent-to-treat (ITT) population, which included all participants who were randomized.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 82 | 163
percentage change | -37.49 (3.866) | -64.52 (2.543)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Squares Mean = -26.97, 95% CI 2-sided [-35.93 to -18.00], Standard Error of Mean 4.572

5. Secondary Outcome: Percentage Change From Baseline in Body Surface Area (BSA) Affected by Psoriasis at Week 16
Description: BSA is a measurement of involved skin of the whole body affected by psoriasis, which ranges from 0% to 100%. Positive percentage change from baseline indicates that a greater BSA was affected by psoriasis. A negative percentage change from baseline indicates that a lesser BSA was affected by psoriasis.
Time Frame: Baseline and Week 16
Population: Measured in the intent-to-treat (ITT) population, which included all participants who were randomized.
Measure: Mean (Standard Error); unit: percentage change in affected BSA
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 82 | 163
percentage change in affected BSA | -20.56 (5.441) | -55.44 (3.428)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Squares Mean = -34.77, 95% CI 2-sided [-46.99 to -22.55], Standard Error of Mean 6.229

6. Secondary Outcome: Percentage of Participants Who Achieved a Children's Dermatology Life Quality Index (CDLQI) Score of 0 or 1 at Week 16
Description: The CDLQI is designed to measure the impact of skin disease on children's quality of life. The CDLQI measures how much the participant's psoriasis has affected them over the last week, and includes 10 questions with possible answers ranging from not at all (score of 0) to very much (score of 3). The CDLQI total score ranged from 0 (no effect on the participant's life) to 30 (extremely large effect on the participant's life). The results presented are for the percentage of participants who achieved a total CDLQI score of 0 or 1 at Week 16.
Time Frame: Week 16
Population: Measured in participants in the intent-to-treat (ITT) population (which included all participants who were randomized), with a baseline CDLQI Score >/= 2.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 76 | 148
percentage of participants | 31.3 | 35.4
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority; p = 0.5616, Cochran-Mantel-Haenszel; Percentage Adjusted Difference = 4.1, 95% CI 2-sided [-9.8 to 18.0]

7. Secondary Outcome: Change From Baseline in CDLQI Score at Week 16
Description: The CDLQI is designed to measure the impact of skin disease on children's quality of life. The CDLQI measures how much the participant's psoriasis has affected them over the last week, and includes 10 questions with possible answers ranging from not at all (score of 0) to very much (score of 3). The CDLQI total score ranged from 0 (no effect on the participant's life) to 30 (extremely large effect on the participant's life). A positive change from baseline score indicates that a participant's quality of life has worsened. A negative change from baseline score indicates that a participant's quality of life has improved.
Time Frame: Baseline and Week 16
Population: Measured in the intent-to-treat (ITT) population, which included all participants who were randomized.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 82 | 163
scores on a scale | -2.7 (0.56) | -5.3 (0.44)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority; p = 0.0009, ANCOVA; Difference in Least Squares Mean = -1.8, 95% CI 2-sided [-2.9 to -0.8]

8. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE) During the Placebo-controlled Phase
Description: An adverse event (AE) was defined as any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of the study. A TEAE is any AE that occurred after first dose of the investigational product.
Time Frame: 16 weeks
Population: Measured in the Safety Population, which included all randomized participants who received at least 1 dose of investigational product. As pre-specified, data are presented per treatment received and adverse event data collected by apremilast dose.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast 20mg; Apremilast 30 mg: In the placebo-controlled phase, participants who were randomized to apremilast who were 20 to < 50 kg received apremilast 20 mg twice daily (BID) for 16 weeks, and participants >/= 50 kg received apremilast 30 mg BID for 16 weeks. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30 mg
Number analyzed (Participants) | 80 | 80 | 83
Participants | 33 | 58 | 48

9. Secondary Outcome: Number of Participants Who Experienced a TEAE During the Apremilast Exposure Period
Description: An AE was defined as any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of the study. A TEAE is any AE that occurred after first dose of the investigational product.
Time Frame: 52 weeks
Population: Measured in the Safety Population, which included all randomized participants who received at least 1 dose of investigational product. As pre-defined in the statistical analysis plan, data are presented per treatment received and adverse event data collected by apremilast dose.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast Exposure Period: Apremilast 20 mg BID: Participants who were randomized to apremilast during the placebo-controlled phase and received apremilast 20 mg BID for 16 weeks during the placebo-controlled phase. At Week 16, participants in the placebo group during the placebo-controlled phase were switched to apremilast 20mg BID for 36 weeks based on baseline weight. Participants who received apremilast 20 mg BID during the placebo-controlled phase continued to receive their original dosing assignment for an additional 36 weeks during the apremilast-extension phase. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Apremilast Exposure Period: Apremilast 30 mg BID: Participants who were randomized to apremilast during the placebo-controlled phase and received apremilast 30 mg BID for 16 weeks during the placebo-controlled phase. At Week 16, participants in the placebo group during the placebo-controlled phase were switched to apremilast 30mg BID for 36 weeks based on baseline weight. Participants who received apremilast 30 mg BID during the placebo-controlled phase continued to receive their original dosing assignment for an additional 36 weeks during the apremilast-extension phase. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
Arm/Group | Apremilast Exposure Period: Apremilast 20 mg BID | Apremilast Exposure Period: Apremilast 30 mg BID
Number analyzed (Participants) | 116 | 119
Participants | 88 | 80

10. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Serious Adverse Event (TESAE) During the Placebo-controlled Phase
Description: A TESAE is any AE occurring at any dose after first dose that results in death, is life-threatening (ie, in the opinion of the Investigator, the participant is at immediate risk of death from the AE), requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay), results in persistent or significant disability/incapacity (a substantial disruption of the participant's ability to conduct normal life functions), is a congenital anomaly/birth defect, or constitutes an important medical event.
Time Frame: 16 weeks
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30 mg
Number analyzed (Participants) | 80 | 80 | 83
Participants | 1 | 2 | 0

11. Secondary Outcome: Number of Participants Who Experienced a TESAE During the Apremilast Exposure Period
Description: as for outcome 10
Time Frame: 52 weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast Exposure Period: Apremilast 20 mg BID | Apremilast Exposure Period: Apremilast 30 mg BID
Number analyzed (Participants) | 116 | 119
Participants | 2 | 1

12. Secondary Outcome: Number of Participants Who Experienced a Treatment-related Adverse Event (TRAE) During the Placebo-controlled Phase
Description: A TREAE is any AE that is determined by the Investigator to have a possibly causal relationship to the investigational product.
Time Frame: 16 weeks
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30 mg
Number analyzed (Participants) | 80 | 80 | 83
Participants | 12 | 36 | 32

13. Secondary Outcome: Number of Participants Who Experienced a TRAE During the Apremilast Exposure Period
Description: as for outcome 12
Time Frame: 52 weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast Exposure Period: Apremilast 20 mg BID | Apremilast Exposure Period: Apremilast 30 mg BID
Number analyzed (Participants) | 116 | 119
Participants | 45 | 47

14. Secondary Outcome: Number of Participants With Diarrhea During the Placebo-controlled Phase
Description: Diarrhea was defined as having 3 or more liquid or watery stools in a day. Participants and their parent/guardian were supplied with diaries (either paper or electronic) that were filled out daily to record and describe any diarrhea and associated symptoms.
Time Frame: Up to approximately 113 days
Population: Measured in participants in the Safety Population (which included all randomized participants who received at least 1 dose of investigational product), who had diary entries at each specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 80 | 163
Participants
  Day 1 to 28: number analyzed (Participants) | 77 | 156
  Day 1 to 28 | 25 | 67
  Day 29 to 56: number analyzed (Participants) | 73 | 155
  Day 29 to 56 | 20 | 51
  Day 57 to 84: number analyzed (Participants) | 73 | 147
  Day 57 to 84 | 14 | 41
  Day 85 to 112: number analyzed (Participants) | 69 | 142
  Day 85 to 112 | 10 | 29
  Day >/= 113: number analyzed (Participants) | 46 | 105
  Day >/= 113 | 2 | 9

15. Secondary Outcome: Number of Participants With Diarrhea During the Apremilast Exposure Period
Description: as for outcome 14
Time Frame: Day 1 up to approximately 365 days
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast Exposure Period: Apremilast 20 mg BID | Apremilast Exposure Period: Apremilast 30 mg BID
Number analyzed (Participants) | 116 | 119
Participants
  Day 1 to 28: number analyzed (Participants) | 109 | 114
  Day 1 to 28 | 36 | 47
  Day 29 to 56: number analyzed (Participants) | 108 | 103
  Day 29 to 56 | 30 | 36
  Day 57 to 84: number analyzed (Participants) | 101 | 110
  Day 57 to 84 | 22 | 32
  Day 85 to 112: number analyzed (Participants) | 100 | 106
  Day 85 to 112 | 17 | 19
  Day 113 to 140: number analyzed (Participants) | 99 | 106
  Day 113 to 140 | 21 | 17
  Day 141 to 168: number analyzed (Participants) | 98 | 104
  Day 141 to 168 | 16 | 21
  Day 169 to 196: number analyzed (Participants) | 96 | 102
  Day 169 to 196 | 19 | 17
  Day 197 to 224: number analyzed (Participants) | 93 | 102
  Day 197 to 224 | 19 | 12
  Day 225 to 252: number analyzed (Participants) | 92 | 98
  Day 225 to 252 | 20 | 12
  Day 253 to 280: number analyzed (Participants) | 76 | 69
  Day 253 to 280 | 18 | 16
  Day 281 to 308: number analyzed (Participants) | 61 | 60
  Day 281 to 308 | 13 | 9
  Day 309 to 336: number analyzed (Participants) | 62 | 59
  Day 309 to 336 | 12 | 5
  Day 337 to 364: number analyzed (Participants) | 59 | 58
  Day 337 to 364 | 7 | 5
  Day >= 365: number analyzed (Participants) | 24 | 22
  Day >= 365 | 1 | 1

16. Secondary Outcome: Number of Participants With Diarrhea Symptoms During the Placebo-controlled Phase
Description: Diarrhea symptoms were nausea, vomiting, abdominal cramps, abdominal pain, fever, bloating, and other symptoms. Participants and their parent/guardian were supplied with diaries (either paper or electronic) that were filled out daily to record and describe any diarrhea and associated symptoms.
Time Frame: Up to approximately 113 days
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 80 | 163
Participants
  Day 1 to 28: number analyzed (Participants) | 77 | 156
  Day 1 to 28: Nausea | 3 | 32
  Day 1 to 28: Vomiting | 2 | 13
  Day 1 to 28: Abdominal cramps | 3 | 16
  Day 1 to 28: Abdominal pain | 9 | 28
  Day 1 to 28: Fever | 1 | 5
  Day 1 to 28: Bloating | 1 | 8
  Day 1 to 28: Other symptoms | 5 | 21
  Day 1 to 28: No symptoms | 53 | 33
  Day 29 to 56: Nausea | 2 | 22
  Day 29 to 56: Vomiting | 2 | 6
  Day 29 to 56: Abdominal cramps | 3 | 7
  Day 29 to 56: Abdominal pain | 9 | 17
  Day 29 to 56: Fever | 0 | 1
  Day 29 to 56: Bloating | 4 | 12
  Day 29 to 56: Other symptoms | 4 | 17
  Day 29 to 56: No symptoms | 56 | 81
  Day 57 to 84: Nausea | 1 | 12
  Day 57 to 84: Vomiting | 0 | 7
  Day 57 to 84: Abdominal cramps | 1 | 9
  Day 57 to 84: Abdominal pain | 5 | 13
  Day 57 to 84: Fever | 0 | 2
  Day 57 to 84: Bloating | 2 | 6
  Day 57 to 84: Other symptoms | 6 | 11
  Day 57 to 84: No symptoms | 65 | 103
  Day 85 to 112: Nausea | 2 | 8
  Day 85 to 112: Vomiting | 1 | 3
  Day 85 to 112: Abdominal cramps | 1 | 5
  Day 85 to 112: Abdominal pain | 2 | 7
  Day 85 to 112: Fever | 0 | 2
  Day 85 to 112: Bloating | 3 | 5
  Day 85 to 112: Other symptoms | 5 | 8
  Day 85 to 112: No symptoms | 66 | 125
  Day >/= 113: Nausea | 0 | 2
  Day >/= 113: Vomiting | 0 | 1
  Day >/= 113: Abdominal cramps | 0 | 1
  Day >/= 113: Abdominal pain | 0 | 2
  Day >/= 113: Fever | 0 | 0
  Day >/= 113: Bloating | 1 | 1
  Day >/= 113: Other symptoms | 0 | 2
  Day >/= 113: No symptoms | 79 | 154

17. Secondary Outcome: Number of Participants With Diarrhea Symptoms During the Apremilast Exposure Period
Description: as for outcome 16
Time Frame: Day 1 up to approximately 365 days
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast Exposure Period: Apremilast 20 mg BID | Apremilast Exposure Period: Apremilast 30 mg BID
Number analyzed (Participants) | 116 | 119
Participants
  Day 1 to 28: number analyzed (Participants) | 109 | 114
  Day 1 to 28: Nausea | 17 | 21
  Day 1 to 28: Vomiting | 10 | 4
  Day 1 to 28: Abdominal cramps | 7 | 9
  Day 1 to 28: Abdominal pain | 21 | 14
  Day 1 to 28: Fever | 2 | 3
  Day 1 to 28: Bloating | 3 | 7
  Day 1 to 28: Other symptoms | 11 | 13
  Day 1 to 28: No symptoms | 38 | 43
  Day 29 to 56: number analyzed (Participants) | 108 | 113
  Day 29 to 56: Nausea | 14 | 10
  Day 29 to 56: Vomiting | 4 | 3
  Day 29 to 56: Abdominal cramps | 4 | 4
  Day 29 to 56: Abdominal pain | 13 | 8
  Day 29 to 56: Fever | 1 | 0
  Day 29 to 56: Bloating | 4 | 9
  Day 29 to 56: Other symptoms | 9 | 9
  Day 29 to 56: No symptoms | 59 | 70
  Day 57 to 84: number analyzed (Participants) | 101 | 110
  Day 57 to 84: Nausea | 6 | 8
  Day 57 to 84: Vomiting | 6 | 4
  Day 57 to 84: Abdominal cramps | 8 | 3
  Day 57 to 84: Abdominal pain | 10 | 6
  Day 57 to 84: Fever | 1 | 1
  Day 57 to 84: Bloating | 1 | 6
  Day 57 to 84: Other symptoms | 10 | 6
  Day 57 to 84: No symptoms | 59 | 76
  Day 85 to 112: number analyzed (Participants) | 100 | 106
  Day 85 to 112: Nausea | 3 | 5
  Day 85 to 112: Vomiting | 3 | 0
  Day 85 to 112: Abdominal cramps | 4 | 2
  Day 85 to 112: Abdominal pain | 6 | 3
  Day 85 to 112: Fever | 1 | 2
  Day 85 to 112: Bloating | 2 | 4
  Day 85 to 112: Other symptoms | 5 | 4
  Day 85 to 112: No symptoms | 76 | 86
  Day 113 to 140: number analyzed (Participants) | 99 | 106
  Day 113 to 140: Nausea | 6 | 2
  Day 113 to 140: Vomiting | 5 | 1
  Day 113 to 140: Abdominal cramps | 4 | 0
  Day 113 to 140: Abdominal pain | 7 | 3
  Day 113 to 140: Fever | 1 | 0
  Day 113 to 140: Bloating | 3 | 2
  Day 113 to 140: Other symptoms | 5 | 3
  Day 113 to 140: No symptoms | 68 | 95
  Day 141 to 168: number analyzed (Participants) | 98 | 104
  Day 141 to 168: Nausea | 5 | 2
  Day 141 to 168: Vomiting | 3 | 1
  Day 141 to 168: Abdominal cramps | 2 | 1
  Day 141 to 168: Abdominal pain | 4 | 2
  Day 141 to 168: Fever | 0 | 0
  Day 141 to 168: Bloating | 2 | 2
  Day 141 to 168: Other symptoms | 3 | 1
  Day 141 to 168: No symptoms | 79 | 95
  Day 169 to 196: number analyzed (Participants) | 96 | 102
  Day 169 to 196: Nausea | 3 | 4
  Day 169 to 196: Vomiting | 2 | 1
  Day 169 to 196: Abdominal cramps | 1 | 2
  Day 169 to 196: Abdominal pain | 7 | 5
  Day 169 to 196: Fever | 0 | 2
  Day 169 to 196: Bloating | 0 | 1
  Day 169 to 196: Other symptoms | 7 | 0
  Day 169 to 196: No symptoms | 76 | 87
  Day 197 to 224: number analyzed (Participants) | 93 | 102
  Day 197 to 224: Nausea | 5 | 2
  Day 197 to 224: Vomiting | 5 | 0
  Day 197 to 224: Abdominal cramps | 1 | 0
  Day 197 to 224: Abdominal pain | 3 | 1
  Day 197 to 224: Fever | 2 | 0
  Day 197 to 224: Bloating | 1 | 1
  Day 197 to 224: Other symptoms | 4 | 1
  Day 197 to 224: No symptoms | 72 | 97
  Day 225 to 252: number analyzed (Participants) | 92 | 98
  Day 225 to 252: Nausea | 9 | 3
  Day 225 to 252: Vomiting | 3 | 0
  Day 225 to 252: Abdominal cramps | 2 | 1
  Day 225 to 252: Abdominal pain | 7 | 1
  Day 225 to 252: Fever | 0 | 0
  Day 225 to 252: Bloating | 3 | 1
  Day 225 to 252: Other symptoms | 4 | 0
  Day 225 to 252: No symptoms | 64 | 92
  Day 253 to 280: number analyzed (Participants) | 76 | 69
  Day 253 to 280: Nausea | 5 | 4
  Day 253 to 280: Vomiting | 1 | 0
  Day 253 to 280: Abdominal cramps | 3 | 1
  Day 253 to 280: Abdominal pain | 6 | 3
  Day 253 to 280: Fever | 1 | 0
  Day 253 to 280: Bloating | 2 | 1
  Day 253 to 280: Other symptoms | 3 | 2
  Day 253 to 280: No symptoms | 55 | 58
  Day 281 to 308: number analyzed (Participants) | 61 | 60
  Day 281 to 308: Nausea | 2 | 3
  Day 281 to 308: Vomiting | 1 | 2
  Day 281 to 308: Abdominal cramps | 1 | 2
  Day 281 to 308: Abdominal pain | 4 | 2
  Day 281 to 308: Fever | 0 | 0
  Day 281 to 308: Bloating | 0 | 1
  Day 281 to 308: Other symptoms | 1 | 1
  Day 281 to 308: No symptoms | 52 | 49
  Day 309 to 336: number analyzed (Participants) | 62 | 59
  Day 309 to 336: Nausea | 2 | 1
  Day 309 to 336: Vomiting | 2 | 0
  Day 309 to 336: Abdominal cramps | 1 | 0
  Day 309 to 336: Abdominal pain | 4 | 0
  Day 309 to 336: Fever | 1 | 0
  Day 309 to 336: Bloating | 1 | 0
  Day 309 to 336: Other symptoms | 4 | 1
  Day 309 to 336: No symptoms | 47 | 57
  Day 337 to 364: number analyzed (Participants) | 59 | 58
  Day 337 to 364: Nausea | 2 | 1
  Day 337 to 364: Vomiting | 1 | 0
  Day 337 to 364: Abdominal cramps | 0 | 0
  Day 337 to 364: Abdominal pain | 2 | 2
  Day 337 to 364: Fever | 0 | 0
  Day 337 to 364: Bloating | 1 | 0
  Day 337 to 364: Other symptoms | 1 | 1
  Day 337 to 364: No symptoms | 52 | 54
  Day >= 365: number analyzed (Participants) | 24 | 22
  Day >= 365: Nausea | 0 | 0
  Day >= 365: Vomiting | 0 | 0
  Day >= 365: Abdominal cramps | 0 | 1
  Day >= 365: Abdominal pain | 0 | 0
  Day >= 365: Fever | 0 | 0
  Day >= 365: Bloating | 0 | 0
  Day >= 365: Other symptoms | 0 | 0
  Day >= 365: No symptoms | 24 | 21

18. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior Per the Columbia-Suicide Severity Rating Scale (C-SSRS) During the Placebo-controlled Phase
Description: The C-SSRS is a questionnaire that is used to assess suicidal ideation and behavior. The C-SSRS questionnaire measures suicidal ideation, intensity of ideation, and suicidal behaviors. Results presented are for the number of participants who recorded suicidal ideation or behavior on the C-SSRS.
Time Frame: 16 weeks
Population: Measured in the Safety Population, which included all randomized participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 80 | 163
Participants | 0 | 0

19. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior Per the C-SSRS During the Apremilast-extension Phase
Description: as for outcome 18
Time Frame: Week 16 to Week 52
Population: Measured in the Safety Population, which included all randomized participants who received at least 1 dose of investigational product who had available C-SSRS data.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast-extension Phase: Apremilast 20 mg BID: At Week 16, participants 20 to < 50 kg received apremilast 20 mg BID for 36 weeks during the apremilast-extension phase. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Apremilast-extension Phase: Apremilast 30 mg BID: At Week 16, participants >/= 50 kg received apremilast 30 mg BID for 36 weeks during the apremilast-extension phase. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
Arm/Group | Apremilast-extension Phase: Apremilast 20 mg BID | Apremilast-extension Phase: Apremilast 30 mg BID
Number analyzed (Participants) | 110 | 111
Participants | 0 | 0

20. Secondary Outcome: Number of Female Participants at Stage I-V of Sexual Development Per Tanner Staging of Sexual Development
Description: The Tanner Staging of sexual development is a scale of physical development as children transition into adolescence and then adulthood. The scale defines physical measurements of development based on characteristics, such as the size of the breasts, genitals, testicular volume, and growth of pubic hair. The scale ranges from stage I (pre-adolescent) to stage V (adult development). The results presented are for the number of participants at stage I-V of development.
Time Frame: Week 52
Population: Measured in the Safety Population, which included all randomized participants who received at least 1 dose of investigational product and had available data for the endpoint. As pre-specified, results are presented based on initial treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 37 | 89
Participants
  Breast Growth: Stage 1 | 8 | 17
  Breast Growth: Stage 2 | 3 | 9
  Breast Growth: Stage 3 | 3 | 9
  Breast Growth: Stage 4 | 6 | 20
  Breast Growth: Stage 5 | 12 | 27
  Breast Growth: Missing | 5 | 7
  Pubic Hair Growth: Stage 1 | 8 | 18
  Pubic Hair Growth: Stage 2 | 3 | 9
  Pubic Hair Growth: Stage 3 | 3 | 9
  Pubic Hair Growth: Stage 4 | 6 | 18
  Pubic Hair Growth: Stage 5 | 12 | 28
  Pubic Hair Growth: Missing | 5 | 7
  Other Changes: Stage 1 | 8 | 18
  Other Changes: Stage 2 | 3 | 9
  Other Changes: Stage 3 | 3 | 12
  Other Changes: Stage 4 | 4 | 16
  Other Changes: Stage 5 | 12 | 26
  Other Changes: Missing | 7 | 8

21. Secondary Outcome: Number of Male Participants at Stage I-V of Sexual Development Per Tanner Staging of Sexual Development
Description: as for outcome 20
Time Frame: Week 52
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 43 | 74
Participants
  Testes Growth: Stage 1 | 11 | 15
  Testes Growth: Stage 2 | 5 | 5
  Testes Growth: Stage 3 | 4 | 10
  Testes Growth: Stage 4 | 5 | 12
  Testes Growth: Stage 5 | 14 | 27
  Testes Growth: Missing | 4 | 5
  Penis Growth: Stage 1 | 11 | 15
  Penis Growth: Stage 2 | 5 | 5
  Penis Growth: Stage 3 | 4 | 11
  Penis Growth: Stage 4 | 5 | 10
  Penis Growth: Stage 5 | 14 | 28
  Penis Growth: Missing | 4 | 5
  Pubic Hair Growth: Stage 1 | 10 | 15
  Pubic Hair Growth: Stage 2 | 5 | 6
  Pubic Hair Growth: Stage 3 | 5 | 8
  Pubic Hair Growth: Stage 4 | 6 | 14
  Pubic Hair Growth: Stage 5 | 13 | 26
  Pubic Hair Growth: Missing | 4 | 5
  Other Changes: Stage 1 | 9 | 15
  Other Changes: Stage 2 | 5 | 5
  Other Changes: Stage 3 | 4 | 8
  Other Changes: Stage 4 | 4 | 11
  Other Changes: Stage 5 | 14 | 26
  Other Changes: Missing | 7 | 9

22. Secondary Outcome: Mean Body Weight of Participants During the Placebo-controlled Phase
Description: The participants' body weight in kilograms (kg) was recorded.
Time Frame: Baseline and Week 16
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 80 | 163
kg
  Baseline | 52.36 (22.177) | 52.04 (21.123)
  Week 16 | 54.18 (22.581) | 51.95 (20.945)

23. Secondary Outcome: Mean Body Weight of Participants During the Apremilast Exposure Period
Description: The participants' body weight in kilograms (kg) was recorded.
Time Frame: Baseline and Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Apremilast Exposure Period: Apremilast 20 mg BID | Apremilast Exposure Period: Apremilast 30 mg BID
Number analyzed (Participants) | 116 | 119
kg
  Baseline | 36.81 (8.954) | 67.94 (19.053)
  Week 52 | 39.04 (9.823) | 67.79 (18.889)

24. Secondary Outcome: Mean Height of Participants During the Placebo-controlled Phase
Description: The participants' height in centimeters (cm) was recorded.
Time Frame: Baseline and Week 16
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 80 | 163
cm
  Baseline | 153.29 (18.435) | 153.33 (18.069)
  Week 16 | 154.54 (17.839) | 154.40 (17.683)

25. Secondary Outcome: Mean Height of Participants During the Apremilast Exposure Period
Description: The participants' height in centimeters (cm) was recorded.
Time Frame: Baseline and Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Apremilast Exposure Period: Apremilast 20 mg BID | Apremilast Exposure Period: Apremilast 30 mg BID
Number analyzed (Participants) | 116 | 119
cm
  Baseline | 140.86 (14.159) | 166.13 (11.416)
  Week 52 | 144.90 (13.944) | 167.84 (10.814)

26. Secondary Outcome: Mean Body Mass Index (BMI) of Participants During the Placebo-controlled Phase
Description: The participants' BMI was calculated as body weight (kg)/height (m^2).
Time Frame: Baseline and Week 16
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 80 | 163
kg/m^2
  Baseline | 21.41 (5.652) | 21.33 (5.197)
  Week 16 | 21.87 (5.883) | 20.98 (5.067)

27. Secondary Outcome: Mean BMI of Participants During the Apremilast Exposure Period
Description: The participants' BMI was calculated as body weight (kg)/height (m^2).
Time Frame: Baseline and Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Apremilast Exposure Period: Apremilast 20 mg BID | Apremilast Exposure Period: Apremilast 30 mg BID
Number analyzed (Participants) | 116 | 119
kg/m^2
  Baseline | 18.32 (2.641) | 24.52 (5.655)
  Week 52 | 18.30 (2.480) | 23.95 (5.539)

28. Secondary Outcome: Number of Participants Who Experienced a Psoriasis Flare During the Placebo-controlled Phase
Description: A psoriasis flare was defined as a sudden intensification of psoriasis (new generalized erythrodermic, inflammatory or pustular psoriasis) requiring medical intervention beyond allowable medications.
Time Frame: 16 weeks
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 80 | 163
Participants | 3 | 2

29. Secondary Outcome: Number of Participants Who Experienced a Psoriasis Flare During the Apremilast Exposure Period
Description: as for outcome 28
Time Frame: 52 weeks
Population: Measured in the Safety Population, which included all randomized participants who received at least 1 dose of investigational product. As pre-defined in the statistical analysis plan, data are presented per treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast Exposure Period: Apremilast 20 mg BID | Apremilast Exposure Period: Apremilast 30 mg BID
Number analyzed (Participants) | 116 | 119
Participants | 7 | 11

30. Secondary Outcome: Number of Participants Who Experienced a Psoriasis Rebound
Description: A psoriasis rebound was defined as an adverse event of psoriasis that started after the last dose date for participants who received treatment in the study.
Time Frame: 14 weeks post last dose (max mean treatment duration in placebo-controlled phase was 15.3 weeks, and 41.9 weeks in the apremilast-exposure period)
Population: Measured in participants in the Safety Population (which included all randomized participants who received at least 1 dose of investigational product) who entered the 14-week observational follow up.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants who received placebo in the placebo-controlled phase who entered the 14-week observational follow up.
- Apremilast 20 mg BID: Participants who received apremilast 20 mg in either the placebo-controlled phase or apremilast extension phase who entered the 14-week observational follow up.
- Apremilast 30 mg BID: Participants who received apremilast 30 mg in either the placebo-controlled phase or apremilast extension phase who entered the 14-week observational follow up.
Arm/Group | Placebo | Apremilast 20 mg BID | Apremilast 30 mg BID
Number analyzed (Participants) | 1 | 14 | 30
Participants | 0 | 0 | 4

ADVERSE EVENTS:
Time Frame: Up to a maximum of 52 weeks
Description: All-cause mortality is reported for all enrolled participants. Serious and other adverse events are reported in the Safety Population, which included all randomized participants who received at least 1 dose of investigational product. As pre-specified, data are presented per treatment received.
Groups:
- Placebo-Controlled Phase: Placebo BID: In the placebo-controlled phase, participants who were randomized to placebo received placebo BID for 16 weeks. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Placebo-Controlled Phase: Apremilast 20 mg BID: In the placebo-controlled phase, participants who were randomized to apremilast who were 20 to < 50 kg received apremilast 20 mg BID for 16 weeks. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Placebo-Controlled Phase: Apremilast 30 mg BID: In the placebo-controlled phase, participants who were randomized to apremilast who were >/= 50 kg received apremilast 30 mg BID for 16 weeks. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Placebo-Controlled Phase: Apremilast BID: In the placebo-controlled phase, participants who were randomized to apremilast who were 20 to < 50 kg received apremilast 20 mg twice daily (BID) for 16 weeks, and participants >/= 50 kg received apremilast 30 mg BID for 16 weeks. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Apremilast Extension Phase: Apremilast 20 mg BID: At Week 16, participants 20 to < 50 kg received apremilast 20 mg BID for 36 weeks. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Apremilast Extension Phase: Apremilast 30 mg BID: At Week 16, participants >/= 50 kg received apremilast 30 mg BID for 36 weeks. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
- Apremilast Extension Phase: Apremilast BID: At Week 16, participants 20 to < 50 kg received apremilast 20 mg BID for 36 weeks, and participants >/= 50 kg received apremilast 30 mg BID for 36 weeks. Participants who completed the study or discontinued the study early could have opted to enter the 14-week observational follow up.
Arm/Group | Placebo-Controlled Phase: Placebo BID | Placebo-Controlled Phase: Apremilast 20 mg BID | Placebo-Controlled Phase: Apremilast 30 mg BID | Placebo-Controlled Phase: Apremilast BID | Apremilast Extension Phase: Apremilast 20 mg BID | Apremilast Extension Phase: Apremilast 30 mg BID | Apremilast Extension Phase: Apremilast BID
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/80 | 0/83 | 0/163 | 0/110 | 0/111 | 0/221
Serious Adverse Events (participants affected / at risk) | 1/80 | 2/80 | 0/83 | 2/163 | 0/110 | 2/111 | 2/221
Other Adverse Events (participants affected / at risk) | 26/80 | 50/80 | 41/83 | 91/163 | 52/110 | 38/111 | 90/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Phase: Placebo BID (N=80) | Placebo-Controlled Phase: Apremilast 20 mg BID (N=80) | Placebo-Controlled Phase: Apremilast 30 mg BID (N=83) | Placebo-Controlled Phase: Apremilast BID (N=163) | Apremilast Extension Phase: Apremilast 20 mg BID (N=110) | Apremilast Extension Phase: Apremilast 30 mg BID (N=111) | Apremilast Extension Phase: Apremilast BID (N=221)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Wandering pacemaker (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Status migrainosus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Testicular appendage torsion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Phase: Placebo BID (N=80) | Placebo-Controlled Phase: Apremilast 20 mg BID (N=80) | Placebo-Controlled Phase: Apremilast 30 mg BID (N=83) | Placebo-Controlled Phase: Apremilast BID (N=163) | Apremilast Extension Phase: Apremilast 20 mg BID (N=110) | Apremilast Extension Phase: Apremilast 30 mg BID (N=111) | Apremilast Extension Phase: Apremilast BID (N=221)
Abdominal pain (Gastrointestinal disorders) | 8 | 23 | 9 | 32 | 14 | 5 | 19
Abdominal pain upper (Gastrointestinal disorders) | 4 | 5 | 4 | 9 | 5 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 8 | 15 | 17 | 32 | 20 | 13 | 33
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 7 | 10 | 2 | 2 | 4
Nausea (Gastrointestinal disorders) | 2 | 15 | 17 | 32 | 18 | 10 | 28
Vomiting (Gastrointestinal disorders) | 2 | 16 | 13 | 29 | 15 | 7 | 22
Pyrexia (General disorders) | 1 | 7 | 3 | 10 | 4 | 1 | 5
COVID-19 (Infections and infestations) | 5 | 2 | 3 | 5 | 4 | 3 | 7
Influenza (Infections and infestations) | 1 | 5 | 2 | 7 | 4 | 2 | 6
Nasopharyngitis (Infections and infestations) | 3 | 5 | 5 | 10 | 8 | 3 | 11
Headache (Nervous system disorders) | 4 | 12 | 5 | 17 | 7 | 5 | 12
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 2 | 5 | 11 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT03701763/Prot_002.pdf
  • Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT03701763/SAP_003.pdf